CLINICAL TRIAL: NCT01692197
Title: A Phase 2 Study of E7070, Idarubicin and Cytarabine in Patients With Relapsed or Refractory Acute Myeloid Leukemia and High-risk Myelodysplastic Syndromes
Brief Title: E7070, Idarubicin and Cytarabine in Relapsed AML and High-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0570; NCI-2012-02065 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; Acute Myelogenous Leukemia; AML; Relapsed or Refractory; High-Risk Myelodysplastic Syndromes; HRMDS; E7070; Idarubicin; Idamycin; Cytarabine; Cytarabine (ARA-C); Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Dexamethasone; Decadron
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Recurrence | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide; Idarubicin; Cytarabine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E7070 + Idarubicin + Cytarabine (Experimental): E7070 400 mg/m2 IV over 1 hour on day 1 and day 8 (+/- 2 days on Day 8 only) followed by, Idarubicin 8 mg/m2 IV over 1 hour daily for 3 days (days 9-11) and Cytarabine 1.0 g/m2 IV over 24 hours daily on day 9-12 (age <60 years) or days 9-11 (age > 60 years). Dexamethasone 10 mg IV daily for 3-4 days with cytarabine.
  Interventions: Drug: E7070; Drug: Idarubicin; Drug: Cytarabine; Drug: Dexamethasone

INTERVENTIONS:
Drug: E7070 — 400 mg/m2 intravenously over 1 hour on Day 1 and Day 8 every 3 weeks.
Drug: Idarubicin — 8 mg/m2 by vein over 1 hour daily for 3 days (Days 9-11).
  Other Names: Idamycin
Drug: Cytarabine — 1.0 g/m2 by vein daily on Days 9 - 12 (age <60 years) or Days 9 - 11 (age > 60 years).
  Other Names: ARA-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Dexamethasone — 10 mg by vein daily for 3 - 4 days with cytarabine.
  Other Names: Decadron

SUMMARY:
The goal of this clinical research study is to learn if E7070 in combination with idarubicin, cytarabine, and dexamethasone can help to control the disease in patients with either AML or high-risk MDS that has relapsed. The safety of the drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

E7070 is designed to stop metabolic ingredients from reaching the cancer cells and to stop the cancer cell from dividing.

Cytarabine is designed to insert itself into DNA (the genetic material of cells) of cancer cells and stop the DNA from repairing itself.

Idarubicin is designed to cause breaks in both strands of DNA (the genetic material of cells).

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body. Dexamethasone is often given to AML patients in combination with other chemotherapy to treat cancer.

Study Drug Administration:

If you are found eligible to take part in this study, you will receive E7070 by vein over 1 hour on Day 1 and Day 8 (+/- 2 days on Day 8 only) followed by idarubicin by vein over 1 hour on Days 9-11. You will also receive cytarabine by vein over 24 hours each day on Days 9-12. If you are 60 years of age or older, you will only receive cytarabine on Days 9-11. On days that you are receiving the cytarabine infusions, you will also receive dexamethasone by vein over about 30 minutes. You will receive dexamethasone before the cytarabine infusions. Each study cycle is about 28 days.

If your doctor thinks you are benefitting from taking the E7070 in combination with idarubicin, cytarabine, and dexamethasone, you may receive up to 2 additional cycles of the study drug combination.

Study Visits:

During Cycle 1, the following tests and procedures will be performed:

* You will be asked about medications you are taking and side effects you may have had.
* Blood (about 2 teaspoons) will be drawn at least 1 time every week for routine tests and to check your liver and kidney function.
* You will have a bone marrow aspirate on Day 28 (+/- 3 days) to check the status of the disease. You may have additional bone marrow aspirates during Cycle 2 if the doctor thinks it is necessary.
* During Cycle 1 only, you will have an ECG on Day 2 (+/- 1 day) and Day 8 (+/- 2 days).

Treatment cycles beyond Cycle 1, the following tests and procedures will be performed:

* You will be asked about medications you are taking and side effects you may have had.
* Blood (about 2 teaspoons) will be drawn every 2-4 weeks for routine tests.
* You will have a bone marrow aspirate to check the status of the disease whenever the doctor feels it is necessary.

Length of Study:

If the doctor thinks you are benefitting with E7070 in combination with idarubicin, cytarabine and dexamethasone, you may receive 2 additional cycles of therapy (a total of 3 cycles on this study.)

You will be taken off study if the disease gets worse, you experience intolerable side effects, or if the study doctor thinks it is in your best interest.

End-of-Treatment Visit:

At the end of treatment, blood (about 2 teaspoons) will be drawn for routine tests within 30 days (+/- 5 days) of your last dose of the study drug combination. You will also be asked about any side effects you may have had.

Long Term Follow-up (unless you have started on alternative therapy):

Blood (about 1 tablespoon) will be drawn for routine tests every 2-3 months for up to 2 years unless the disease gets worse or you start on another treatment.

This is an investigational study. E7070 is not FDA-approved or commercially available for use in patients with AML or MDS that has relapsed. Its use in this study is considered investigational. Idarubicin, cytarabine, and dexamethasone are FDA-approved and commercially available for use in the treatment of AML. The combination of E7070, idarubicin, cytarabine, and dexamethasone in this study is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with histologically or cytologically confirmed relapsed or refractory acute myeloid leukemia (AML) [except acute promyelocytic leukemia], or high-risk myelodysplastic syndrome (HRMDS) (Int-2 high risk by International Prostate Symptom Score (IPSS) or >10% blasts in marrow).
2. Patients must be 18 years or older.
3. Patients must have a performance status of 0-2 (Zubrod scale).
4. Patients must have adequate renal function (serum creatinine less than or equal to 1.3 mg/dL and/or creatinine clearance > 40 mL/min). Patients with renal dysfunction due to organ infiltration by disease may be eligible after discussion with the Principal Investigator (PI) (up to creatinine less than or equal to 2.0), and appropriate dose adjustments will be considered.
5. Patients must have adequate hepatic function (bilirubin less than or equal to 2.0 mg/dl; SGOT or Serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 times the ULN for the reference lab unless due to leukemia or congenital hemolytic disorder or bilirubin). Patients with hepatic dysfunction (SGOT/SGPT up to less than or equal to 5 X ULN) due to organ infiltration by disease may be eligible after discussion with the PI, and appropriate dose adjustments will be considered.
6. Patients must have normal cardiac ejection fraction
7. QTc interval </= 480 msecs.
8. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
9. Female patients must not be pregnant or lactating. Female patients of childbearing potential (including those <1 year post-menopausal) and male patients must agree to use contraception.

Exclusion Criteria:

1. Patients must not have untreated or uncontrolled life-threatening infection.
2. Patients must not have received chemotherapy and/or radiation therapy within 2 weeks. Hydroxyurea is allowed up to 48 hours prior to starting therapy in the setting of rapidly proliferating disease. Use of hydroxyurea to control proliferative disease will be allowed starting from day 2 until day 7 Cycle 1. Maximum dose of hydroxyurea allowed daily is 5 gram and hydroxyurea must be discontinued once administration of idarubicin and cytarabine is started.
3. Any other medical condition, including mental illness or substance abuse, deemed by the PI to be likely to interfere with a patient's ability to sign informed consent or cooperate and participate in the study or with the interpretation of the results.
4. Patients must not have received an investigational anti-cancer drug within two weeks of E7070 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2/2013 to 06/2014
Pre-assignment Details: Of the 43 participants registered, three never received the study medication.
Groups:
- E7070 and Idarubicin and Cytarabine: E7070 400 mg/m2 intravenously (IV) approximately over 1 hour on day 1 and day 8:
  Idarubicin 8 mg/m2 IV approximately over 1 hour daily x 3 (days 9-11) Cytarabine 1.0 g/m2 IV approximately over 24 hours daily on day 9-12 (age <60 years) or days 9-11 (age ≥ 60 years).
  Dexamethasone 10 mg IV daily for 3-4 days with cytarabine (Duration is approximately 28 days).
Period: Overall Study
Arm/Group | E7070 and Idarubicin and Cytarabine
Started | 43
Completed | 40
Not Completed | 3
Not completed — Failed Screening | 3

BASELINE CHARACTERISTICS:
Arm/Group | E7070 and Idarubicin and Cytarabine
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 63 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Efficacy measured by overall response - complete response plus complete response with incomplete platelet recovery, plus partial response (Complete remission (CR) + Complete remission without platelet recovery (CRp) + Partial Remission (PR)+ marrow clearance of blast) during cycle 1.
Time Frame: 2 cycles (60 days)
Population: Thirty seven patients are evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | E7070 and Idarubicin and Cytarabine
Number analyzed (Participants) | 37
Participants | 11

2. Secondary Outcome: Disease-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 5 years
Population: Thirty seven patients are evaluable.
Measure: Median (Full Range); unit: months
Arm/Group | E7070 + Idarubicin + Cytarabine
Number analyzed (Participants) | 37
months | 1.7 [1 to 42]

3. Secondary Outcome: Duration of Response
Description: Response date to loss of response or last follow up.
Time Frame: Up to 5 years
Population: Thirty seven patients are evaluable.
Measure: Median (Full Range); unit: months
Arm/Group | E7070 and Idarubicin and Cytarabine
Number analyzed (Participants) | 37
months | 6.7 [1 to 13]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last follow-up.
Time Frame: Up to 5 years
Population: Thirty seven patients are evaluable.
Measure: Median (Full Range); unit: months
Arm/Group | E7070 and Idarubicin and Cytarabine
Number analyzed (Participants) | 37
months | 5.1 [1 to 42]

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected beginning from the time the subject signs the study consent until resolution or for 30 days after the participants last study visit.
Arm/Group | E7070 and Idarubicin and Cytarabine
All-Cause Mortality (participants affected / at risk) | 11/40
Serious Adverse Events (participants affected / at risk) | 30/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E7070 and Idarubicin and Cytarabine (N=40)
Allergic Reaction (General disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (2)
Back Pain (General disorders) | 1 (1)
Bone Marrow Hypocellular (General disorders) | 1 (1)
Bone Pain (General disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Death (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infective Endocarditis (Infections and infestations) | 1 (1)
Fall (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 14 (18)
Fever (General disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Hypotension (Cardiac disorders) | 1 (1)
Injection Site Reaction (Investigations) | 1 (1)
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Joint Infection (Infections and infestations) | 1 (2)
Lung Infection (Infections and infestations) | 11 (15)
Multi-Organ Failure (General disorders) | 1 (1)
Pelvic Infection (Infections and infestations) | 1 (1)
Pulmonary edema (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 9 (10)
Skin Infection (Infections and infestations) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E7070 and Idarubicin and Cytarabine (N=40)
Pain (General disorders) | 6 (7)
Acute Kidney injury (Renal and urinary disorders) | 2 (2)
Agitation (Nervous system disorders) | 2 (2)
Increased Alanine Aminotransferase (Metabolism and nutrition disorders) | 9 (15)
Increased Alkaline Phosphatase (Metabolism and nutrition disorders) | 6 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 11 (11)
Anxiety (Nervous system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Increased Aspartate Aminotransferase (Metabolism and nutrition disorders) | 8 (11)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 14 (28)
Increased Cardiac Troponin I (Cardiac disorders) | 2 (2)
Chest Pain (Cardiac disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Confusion (Nervous system disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 13 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Increased Creatinine (Metabolism and nutrition disorders) | 9 (12)
Dehydration (Gastrointestinal disorders) | 3 (3)
Depression (Nervous system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 17 (17)
Dizziness (General disorders) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Edema (Blood and lymphatic system disorders) | 14 (16)
Epistaxis (Blood and lymphatic system disorders) | 3 (3)
Eye Disorders (Eye disorders) | 2 (2)
Fatigue (General disorders) | 16 (17)
Neutropenic Fever (Infections and infestations) | 10 (13)
Fever (General disorders) | 8 (10)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (11)
Hallucinations (Nervous system disorders) | 3 (3)
Headache (General disorders) | 7 (8)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Hiccups (Gastrointestinal disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (29)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Cardiac disorders) | 2 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (33)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (23)
Hypokalemia (Metabolism and nutrition disorders) | 17 (33)
Hypomagnesemia (Metabolism and nutrition disorders) | 16 (20)
Hyponatremia (Metabolism and nutrition disorders) | 10 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (20)
Hypotension (Cardiac disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Insomnia (General disorders) | 6 (6)
Lethargy (General disorders) | 2 (2)
malaise (General disorders) | 3 (3)
Oral Mucositis (Gastrointestinal disorders) | 3 (3)
Nasal Congestion (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 21 (26)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sinus Tachycardia (Cardiac disorders) | 5 (5)
Skin and Subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 13 (14)
Sore Throat (Gastrointestinal disorders) | 2 (2)
Surgical and Medical Procedures (Surgical and medical procedures) | 3 (3)
Urinary Retention (Renal and urinary disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 9 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT01692197/Prot_SAP_000.pdf